CLINICAL TRIAL: NCT05083832
Title: Effects of Ultrasound-guided Continuous Erector Spina Plane Block and Continuous Serratus Anterior Plane Block on Post-thoracotomy Pain
Brief Title: Effect of Two Different Plane Blocks on Post-thoracotomy Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atatürk Chest Diseases and Chest Surgery Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Musa Zengin, Principal İnvestigator, Atatürk Chest Diseases and Chest Surgery Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E.Kurul-E1-21-1863
Record Dates: First submitted 2021-10-06; First posted 2021-10-19 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Pain, Postoperative; Thoracotomy; Erector Spinae Plane Block; Serratus Anterior Plane Block
Keywords: Pain, Postoperative; Thoracotomy; Erector spinae plane block; Serratus anterior plane block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous erector spinae plane block (Active Comparator): Following the visualization of the anatomical structures, the nerve block needle was advanced via the in-plane technique beneath the erector spinae muscles until the interfascial space was reached. After hydrodissection with 2 ml normal saline, 20 ml 0.25% bupivacaine was injected into the area. A catheter will be placed in this area. Then, 5 ml/hour 0.125% bupivacaine will be infused via erector spinae plane block catheter.
  Interventions: Procedure: Continuous Erector Spina Plane Block vs Continuous Serratus Anterior Plane Block
- Continuous serratus anterior plane block (Active Comparator): Following the visualization of the anatomical structures, the nerve block needle was advanced via the in-plane technique beneath the serratus anterior muscles until the fourth rib area. After hydrodissection with 2 ml normal saline, 20 ml 0.25% bupivacaine was injected into the area. A catheter will be placed in this area. Then, 5 ml/hour 0.125% bupivacaine will be infused via serratus anterior plane block catheter.
  Interventions: Procedure: Continuous Erector Spina Plane Block vs Continuous Serratus Anterior Plane Block

INTERVENTIONS:
Procedure: Continuous Erector Spina Plane Block vs Continuous Serratus Anterior Plane Block — Two different catheter techniques with same doses local anesthetic infusion

SUMMARY:
Thoracotomy is recognized as one of the most painful surgical procedures. This increases the frequency of postoperative pulmonary complications. Erector Spinae Plane Block (ESPB) and Serratus Anterior Plane Block (SAPB) are more superficial, easier to perform, and less likely to have complications. In addition, ESPB and SAPB applications are increasing in patients who underwent thoracotomy and thoracoscopic surgery.

In this study, the investigators aimed to evaluate the effect of continuous ESPB and continuous SAPB via US-guidance on post-thoracotomy pain.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years old
* ASA physical status I-II-III
* BMI 18 to 30 kg/m2
* Elective thoracotomy surgery

Exclusion Criteria:

* Patient refusing the procedure
* Emergency surgery
* History of chronic opioid or analgesic used

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Pain scores | 72 hours after surgery
  Pain will be assessed at rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain). Pain assessment will be done at 1st, 2nd, 4th, 8th, 16th, 24th, 48th and 72nd hours after surgery.

SECONDARY OUTCOMES:
Morphine consumption | 24 hours after surgery
  Morphine consumption for 24 hours will be recorded
Side effects | 72 hours after surgery
  Side effects, such as allergy to local anesthetics, hypotension, nausea/vomiting, itching, headache, and sweating will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Atatürk Chest Disease and Chest Surgery Training and Research Hospital, Keçiören, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No